CLINICAL TRIAL: NCT06643234
Title: Sublay Versus Intraperitoneal Onlay Mesh Repair in Large Ventral Hernias. A New Technique
Brief Title: Sublay Versus Intraperitoneal Onlay Mesh Repair in Large Ventral Hernias
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Kahlawy Mahrous Mohamed (Other)
Responsible Party: Sponsor-Investigator, Ahmed Kahlawy Mahrous Mohamed, Principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Large abdominal hernia
Record Dates: First submitted 2024-09-29; First posted 2024-10-16 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) modified sublay hernioplasty: (Active Comparator): In the classic sublay hernioplasty technique, the hernia sac remains unopened. The procedure involves dissection of the posterior rectus sheath, which is then sutured at the midline. A mesh is placed behind the rectus muscle and in front of the posterior rectus sheath. Subsequently, the rectus muscle and anterior rectus sheath are sutured together at the midline, introducing tension to the repair. Conversely, the modified sublay hernioplasty technique follows a similar approach but with a key difference: the rectus muscle and anterior rectus sheath are left undisturbed without suturing them together. This modification aims to achieve a tension free repair, potentially reducing complications and enhancing overall outcomes.
  Interventions: Procedure: Ventral hernia repair
- Group (B) IPOM: (Active Comparator): The hernia repair procedure involved several key steps. First, the hernial sac was fully exposed and completely removed. Following this, a synthetic mesh was placed internally, covering the defect with overlapping edges to ensure adequate reinforcement. The mesh was then fixed to the anterior abdominal wall using sutures, which were applied through the supporting layers of the abdominal wall to secure the mesh in place. Preoperatively, all patients underwent comprehensive general and local examinations, routine laboratory blood tests, and abdominal ultrasound to evaluate the size of the hernia defect.
  Interventions: Procedure: Ventral hernia repair

INTERVENTIONS:
Procedure: Ventral hernia repair — Comparative between both techniques

SUMMARY:
The aims of this study is to compare the efficacy of modified sublay hernioplasty versus intraperitoneal onlay mesh repair for large ventral hernias.

Specifically, this study will assess the primary outcome of recurrence rate one year post surgery and evaluate secondary outcomes, including intraoperative complications, infection rates, pain levels, and post operative hospital stay durations.

DETAILED DESCRIPTION:
In general surgery, the management of ventral abdominal hernias characterized by the protrusion of tissue through weaknesses in the abdominal wall presents significant challenges, particularly when dealing with large ventral hernias, defined as those ≥10 cm or those under tension if closed primarily.

Incisional hernias, a specific subset of ventral hernias, add to the complexity of repair.

While the Intraperitoneal Onlay Mesh (IPOM) technique is noted for its reduced surgical and postoperative complications and lower reoperation rates, it also suffers from high costs, limited availability of specialized meshes like dynamesh, and increased intraoperative complications.

Alternatively, the modified open sublay technique, which employs a primary retro-muscular fascial repair and uses an affordable polypropylene mesh, offers a promising and cost effective solution with potential for a tension free repair.

This thesis aims to evaluate and compare these techniques to identify the most effective approach for large ventral hernia repair, balancing surgical outcomes, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-70) years, both sexes.
* Fitness for surgery.
* Patients with uncomplicated ventral hernia.
* Large anterior abdominal wall defect.

Exclusion Criteria:

* Patients don't fit for general anesthesia due to sever co-morbidity.
* Patients with complicated ventral hernia.
* Patient refusal of surgical intervention.
* History of bleeding disorders.
* Pregnancy in female patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
-Recurrence rate one year post operative. | 1 year postoperative
  Number of recurrent cases

SECONDARY OUTCOMES:
1-infection rates(number of cases) 2-pain level( according to Visual Analog Score for pain) 3-post operative hospital stay duration(number of days) 4-intra and post operative complications(as iatrogenic injury and adhesions). | 1 year postoperative
  The number of cases come with post operative infection , pain(according to pain rating scale) , postoperative days of stay and intraoperative complications.

REFERENCES:
- [Background] Kockerling F, Simon T, Adolf D, Kockerling D, Mayer F, Reinpold W, Weyhe D, Bittner R. Laparoscopic IPOM versus open sublay technique for elective incisional hernia repair: a registry-based, propensity score-matched comparison of 9907 patients. Surg Endosc. 2019 Oct;33(10):3361-3369. doi: 10.1007/s00464-018-06629-2. Epub 2019 Jan 2. PMID 30604264